CLINICAL TRIAL: NCT01987154
Title: Tolerance of an Extensively Hydrolyzed Protein Infant Formula Versus a Premature Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 6020
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Feeding Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed cow milk-based premature infant formula (Active Comparator)
  Interventions: Other: Marketed cow milk-based premature infant formula
- Marketed extensively hydrolyzed casein infant formula (Experimental)
  Interventions: Other: Marketed extensively hydrolyzed casein infant formula

INTERVENTIONS:
Other: Marketed cow milk-based premature infant formula
  Arms: Marketed cow milk-based premature infant formula
Other: Marketed extensively hydrolyzed casein infant formula
  Arms: Marketed extensively hydrolyzed casein infant formula

SUMMARY:
To evaluate the use of a hypoallergenic infant formula containing an extensively hydrolyzed protein source for routine nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant 28 to 33 weeks gestational age, inclusive, at birth
* Infant has never received enteral feedings or current enteral intake is less than 30 mL/kg/day
* Birth weight is greater than or equal to 700g to 1750g
* Appropriate birth weight for gestational age
* Singleton or twin birth
* Signed Informed consent

Exclusion Criteria:

* Infant's mother plans to exclusively breast feed
* 5 minute APGAR score is less than or equal to 4
* Major surgery that required general anesthesia prior to randomization
* Ventilator-dependent or requiring greater than 40% FiO2 on day of randomization
* Grade III or IV intraventricular hemorrhage diagnosed prior to randomization
* Infant is currently participating in another clinical study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Enteral intake (ml/kg/day) | Daily for 14 days

SECONDARY OUTCOMES:
Body Weight (g) | Daily for 14 days
Feeding Tolerance | Daily for 14 days
  Gastric residuals, regurgitation(>1 ml), fecal output (number of stools per day)
Respiratory status | Daily for 14 days
  Apnea and/or bradycardia events, use of supplemental oxygen, use of mechanical ventilation
Gut Inflammation | Once at Study Day 14
  Fecal calprotectin, alpha and beta defensins, TNF alpha, gastric ultrasound
Confirmed or suspected sepsis or necrotizing enterocolitis | Daily for 14 days
Date of hospital discharge | Once at hospital discharge
Growth | Study Days 1, 7, and 14
  length (cm) and head circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Mariella Baldassarre, M.D., Principal Investigator — Universita degli Studi di Bari
Locations (1):
- Azienda Ospedaliera "Ospedale Policlinico Consorziale" di Bari, Bari, Apulia, Italy